CLINICAL TRIAL: NCT07031297
Title: Upper Body Subcutaneous Adipose Tissue Outflow Response to a Meal
Brief Title: Upper Body Subcutaneous Exosome Release in Response to a Meal in Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kelli A. Lytle, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24-007465
Record Dates: First submitted 2025-05-23; First posted 2025-06-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal weight group (Other): 5 male and 5 female volunteers in normal weight range
  Interventions: Diagnostic Test: Meal Study
- Obesity group (Other): 5 male and 5 female volunteers with obesity (BMI 29.0-35.0 kg/m2)
  Interventions: Diagnostic Test: Meal Study

INTERVENTIONS:
Diagnostic Test: Meal Study — Participants will consume a mixed meal drink (Ensure) equivalent to 40% of basil metabolic rate as calculated via Harris Benedict equation.
  Following consumption of the drink they will undergo a series of blood draws over the following 4 hours:
  * Plasma glucose will be measured according to a mixed meal test protocol every 10 minutes for the first hour and then every 15, then 30 minutes for the last 3 hours.
  * 1 ml plasma aliquots for exosome analysis and insulin concentrations will be drawn every 30 minutes following consumption of ensure for 4 hours.
  * Blood gasses will be drawn every 30 minutes for the 4 hours following the meal.
  Participants will undergo a second abdominal adipose tissue biopsy 3 hours following mixed meal drink.

SUMMARY:
The purpose of this study is to understand the specific outflow and difference between normal weight and volunteers with obesity of upper body subcutaneous adipose tissue in response to a mixed meal challenge by site specific cannulation of the superior epigastric vein. We will characterize the exosome signatures in response to a meal and compare to the exosome signature of arterialized venous plasma samples.

ELIGIBILITY:
Inclusion Criteria:

• All women must be premenopausal

Exclusion Criteria:

* Participants taking medications know to affect blood flow (statins, β-blockers) or fatty acid or adipose tissue metabolism (TZDs, high dose fish oil supplements)
* Diabetes, history of cardiovascular disease
* Allergy to lidocaine
* Post-menopausal women
* Pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Adipose tissue blood flow | 4 hours
  Blood flow will be measured in the upper body subcutaneous adipose tissue using Xenon washout and reported as blood flow in ml/min/100g adipose tissue.

SECONDARY OUTCOMES:
Glucose | Baseline, 4 hours
  Sugar in the form of glucose in the blood. The concentration of glucose in the blood. A healthy normal range is 70 to 99 mg/dL, results reported in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Kelli A Lytle, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No